CLINICAL TRIAL: NCT03300089
Title: Effect of Anaesthetic Techniques on Clinical Outcome After Lumbar Spine Surgery: Regional Versus General Anaesthesia. A Prospective Randomized Controlled Trial
Brief Title: Lumbar Spine Surgery: Regional vs. General Anaesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Anna Clinic Luzern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EKNZ 2015-261
Record Dates: First submitted 2017-09-27; First posted 2017-10-03 (Actual); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Herniated Disk Lumbar
MeSH Terms: interventions — Anesthesia, General; Anesthesia, Conduction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes Assessor and statistician are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General Anaesthesia (Active Comparator): General Anaesthesia during surgery
  Interventions: Procedure: General anaesthesia
- Regional Anaesthesia (Experimental): Regional Anaesthesia during surgery
  Interventions: Procedure: Regional anaesthesia

INTERVENTIONS:
Procedure: General anaesthesia — General anaesthesia
  Arms: General Anaesthesia
Procedure: Regional anaesthesia — Regional anaesthesia
  Arms: Regional Anaesthesia

SUMMARY:
Background: Lumbar spine surgery can be performed using different anaesthetic techniques such as general endotracheal anaesthesia (GA) or spinal-based regional anaesthesia (RA), that have different side effect profiles (e.g. opioids - nausea, vomiting, pruritus, sedation; local anaesthetics - motor weakness) which may affect quality of recovery in different ways.

Aim of the study: The purpose of this study is to determine the effects of GA and RA in lumbar spine surgery on clinical outcome, combining validated patient-reporting instruments and morbidity such as serious adverse events.

Hypothesis: The investigators hypothesize that in patients undergoing lumbar spine surgery, RA shows significant advantages as compared to GA with respect to the postoperative pain score, the degree of postoperative nausea and vomiting (PONV), the postoperative anaesthetic care unit (PACU) and anaesthesia time and the satisfaction of patients and surgeons.

Design of the study: This is a single-centre two-arm randomised-controlled trail.

DETAILED DESCRIPTION:
1. Background Lumbar spine surgery can be performed using different anaesthetic techniques such as general endotracheal anaesthesia (GA) or spinal-based regional anaesthesia (RA). In a recent review several studies showed a decreased postoperative pain score in the RA groups (1). But only few randomized control trials (RCT) have been performed comparing these two anaesthetic techniques and have shown partly conflicting results (2-5).

   Each anaesthetic agent or regimen has a particular side effect profile (e.g. opioids - nausea, vomiting, pruritus, sedation; local anaesthetics - motor weakness) which may affect quality of recovery in different ways. Although there are few data examining the correlation between side effects from different analgesic regimens and quality of recovery per se, some data suggest different analgesic regimens will result in different side effects and consequently different levels of quality of recovery.

   Although inconsistent data exist covering surgery time, anaesthesia time, postoperative anaesthetic care unit (PACU) time and postoperative analgesic dose requirements (6-8).

   But there are some hinds that RA leads to better results concerning postoperative mortality and morbidity in opposite to general anaesthesia (9-10). Also RA showed better results concerning economic aspects (11,12).

   No clinical trials have sufficient subject numbers to determine definitively the effects of anaesthetic techniques on minor or major benefits concerning clinical outcome. There is insufficient evidence to confirm or deny the ability of these two anaesthetic techniques to affect major postoperative mortality or morbidity and there is currently no sufficient evidence that RA or GA have any clinically significant beneficial effect on postoperative outcome. Further there are still insufficient data to determine if the type of anaesthetic technique, degree of analgesia and the presence of side effects may influence quality of life, quality of recovery, patient and surgeon's satisfaction and length of hospitalisation.

   There are few data examining the correlation between side effects from different anaesthetic regimens and quality of recovery per se, some data suggest different analgesic regimens may result in different side effects and consequently different levels of quality of recovery.

   Although there are data suggesting that improved postoperative analgesia leads to better patient outcomes, there is insufficient evidence to support subsequent improvements inpatient-centered outcomes such as quality of life and quality of recovery. So the correlation between RA and different outcome parameters are very complex and up to now there is no clear evidence for any recommendation concerning the use of RA or GA in generally (13).
2. Study Objective Lumbar spine surgery can be performed using different anaesthetic techniques such as general endotracheal anaesthesia (GA) or spinal-based regional anaesthesia (RA). The purpose of this study is to determine the effects of two different anaesthetic techniques and their impact on clinical outcome.

   Further this study is developed to combine validated patient-reported instruments with the assessment of the effect of different anaesthetic techniques on patient-reported outcomes in the peri-and postoperative period.
3. Hypothesis The investigators hypothesize that for patients undergoing lumbar spine surgery, the performing of a RA shows significant benefits in comparison with patients receiving GA. It concerns the postoperative pain score, the degree of PONV, the PACU and anaesthesia time and the patient's and surgeons's satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patient must give informed consent before registration.
* Age ≥ 18 years
* Physical Status Classification of the American Society of Anaesthesiologists Score (ASA) ≤ 3
* Patient with a diagnosed lumbar spinal stenosis or a herniated lumbar disc for elective neurosurgery

Exclusion Criteria:

* ASA ≥ 4
* Infection at the site of the operation field
* Longterm History (≥ 6 month) of neuropathic pain on the operation site
* Revision surgery and/or follow-up operations
* Severe coagulopathy (platelet count < 100.000 / mL3 or Thromboplastin time < 50%)
* Allergy to local anaesthetics or opioids
* Previous drug dependency or chronic use of opioids (≥ 6 month)
* Psychiatric disorder precluding understanding of information on trial related topics or given informant consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-01-19 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-07-20 (Actual)

PRIMARY OUTCOMES:
Morphine consumption | From immediately after the operation until 48 hours postoperative
  Cumulated morphine consumption in mg

SECONDARY OUTCOMES:
VAS score | Postoperative at the day of surgery until 48 hours postoperative
  Visual Analog Pain assessment, assessed each day
Anesthesia time | Day of surgery
  Duration of anesthesia in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Bertram Bänziger, MD, Principal Investigator — Klinik St. Anna Luzern
Locations (1):
- St. Anna Hospital, Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] De Rojas JO, Syre P, Welch WC. Regional anesthesia versus general anesthesia for surgery on the lumbar spine: a review of the modern literature. Clin Neurol Neurosurg. 2014 Apr;119:39-43. doi: 10.1016/j.clineuro.2014.01.016. Epub 2014 Jan 27. PMID 24635923